CLINICAL TRIAL: NCT05114941
Title: A Prospective, Multi-center, Randomized Parallel Controlled Clinical Study on the Efficacy and Safety of Protein A Immunoadsorption and Intravenous Immunoglobulin in the Treatment of Guillain-Barre Syndrome
Brief Title: Comparison of the Efficacy and Safety of Immunoadsorption and Intravenous Immunoglobulin for Guillain-Barre Syndrome
Acronym: GBS-PRAISING
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Wang Miao, professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-KY-0709
Record Dates: First submitted 2021-10-21; First posted 2021-11-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Guillain-Barre Syndrome
Keywords: immunoadsorption; intravenous immunoglobulin
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunoadsorption group (Experimental): Protein A immunoadsorption therapy
  Interventions: Device: immunosorbent column
- intravenous immunoglobulin group (Active Comparator): Treatment with intravenous immunoglobulin
  Interventions: Drug: intravenous immunoglobulin

INTERVENTIONS:
Device: immunosorbent column — Immunoadsorption treatment regimen: the treatment is performed once every 1-3 days, at least 5 times, and the amount of regenerated plasma for each treatment is 1 to 3 times the plasma volume. The immunosorbent column adopts the protein A immunosorbent column.
  Other Names: Protein A Immunoadsorption
  Arms: Immunoadsorption group
Drug: intravenous immunoglobulin — Intravenous immunoglobulin treatment regimen: intravenous immunoglobulin therapy, 400mg/kg/d, once a day, for at least 5 consecutive days.
  Arms: intravenous immunoglobulin group

SUMMARY:
Guillain-Barre syndrome is an immune-mediated acute inflammatory peripheral neuropathy. The currently effective treatment methods include intravenous immunoglobulin and plasma exchange. Immunoadsorption has been widely used to treat immune-related diseases. There are currently no prospective large-sample clinical trials of immunoadsorption therapy for Guillain-Barre syndrome. The neuro-intensive care unit of the First Affiliated Hospital of Zhengzhou University is preparing to carry out a prospective, multi-center, randomized parallel controlled clinical study on the efficacy and safety of protein A immunoadsorption and intravenous immunoglobulin (IVIG) in the treatment of Guillain-Barre syndrome. It is estimated that 204 patients with Guillain-Barre syndrome will be included. The patients will be randomly assigned to the immunoadsorption group and the IVIG group. The primary outcome measure: changes in Hughes scores (4 weeks after starting treatment vs. baseline (before starting treatment) ). This study aims to explore the efficacy and safety of protein A immunoadsorption and intravenous immunoglobulin in the treatment of Guillain-Barre syndrome.

DETAILED DESCRIPTION:
Guillain-Barre syndrome (GBS) is an immune-mediated acute inflammatory peripheral neuropathy. The currently proven effective treatment methods include intravenous immunoglobulin and plasma exchange. In the clinical treatment process, the plasma source is often stressed, forcing the treatment to be terminated. Intravenous immunoglobulin therapy may cause allergies. Based on the above reasons, immunosorbent technology came into being.

Immunoadsorption technology is widely used in clinical treatment of immune-related diseases. Protein A can recognize and bind to the Fc segment of human antibodies. The protein A immunosorbent column uses recombinant staphylococcal protein A as its ligand. The protein can specifically recognize and bind to the Fc segment of human antibodies, so it can adsorb human antibodies, mainly immunoglobulin G, and can adsorb immunoglobulin M and immunoglobulin A at the same time. The binding of protein A and antibody is reversible.

Immunoadsorption therapy has obvious advantages: The patient's own plasma is transfused without replacement fluid; It can prevent infection Diseases such as viral hepatitis, AIDS, etc.; The adsorption is selective or specific, and normal plasma components including coagulation factors, etc., only slightly decrease; Does not affect the simultaneous drug treatment; The protein A immunosorbent column can be reused; The treatment effect is better, and the amount of plasma purified by a single immunoadsorption is 1.5 to 3 times that of plasma exchange.

The First Affiliated Hospital of Zhengzhou University is preparing to carry out a prospective, multi-center, randomized parallel controlled clinical study on the effectiveness and safety of protein A immunoadsorption and intravenous immunoglobulin in the treatment of Guillain-Barre syndrome. The control group received intravenous immunoglobulin injections using the standard treatment recommended by the Guilan-Barre Syndrome Guidelines. Compare the effectiveness and safety of the two treatment regimens in the treatment of Guillain-Barre syndrome, and explore a more effective and safe treatment regimen for the treatment of Guillain-Barre syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of Guillain - Barre syndrome;
2. The onset is within 2 weeks;
3. Age is greater than or equal to 18 years old and less than or equal to 60 years old;
4. Hughes function classification is greater than or equal to 3;
5. The subject or his legal representative can understand the purpose of the research, show sufficient compliance with the research protocol, and sign an informed consent form.

Exclusion Criteria:

1. Those who are pregnant;
2. Three months before the screening period, receive immunoadsorption therapy or intravenous immunoglobulin therapy;
3. Those who have a history of allergies in the membrane of the plasma separator;
4. Those who must use angiotensin-converting enzyme inhibitor drugs within 1 week before being included in the trial and during treatment and cannot be stopped;
5. Severe active bleeding or diffuse intravascular coagulation, patients with systemic circulatory failure that are difficult to correct with drugs;
6. Severe cardiac insufficiency, that is, those who have reached NYHA IV according to the heart failure classification standards of the New York Heart Association (NYHA);
7. There are contraindications to intravenous immunoglobulin;
8. Those with other system autoimmune diseases;
9. Diagnosis of variant GBS: such as Miller-Fisher syndrome, GBS with cranial nerve damage, sensory GBS, pan-autonomous GBS. Patients with chronic inflammatory demyelinating polyperipheral neuropathy whose condition has been significantly alleviated when visiting a doctor;
10. Subjects who have participated in any other drug or medical device clinical trials within 1 month before entering the screening period; Note: Subjects who participated in observational studies (that is, the study does not require changes or other interventions) will not be excluded;
11. Patients who cannot obtain informed consent;
12. Those who cannot receive active and comprehensive treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Hughes scores | 4 weeks after starting treatment vs. baseline (before starting treatment)
  Compared with the patient's Hughes score before treatment, the change of Hughes scores 4 weeks after the start of protein A immunoadsorption or intravenous immunoglobulin treatment.

SECONDARY OUTCOMES:
Changes in Hughes scores | 2 weeks after starting treatment vs. baseline (before starting treatment)
  Compared with the patient's Hughes score before treatment, the change of Hughes scores 2 weeks after the start of protein A immunoadsorption or intravenous immunoglobulin treatment.
Reached Hughes Grade 2 | From date of first treatment until the date of patient's recovery to Hughes Grade 2 or end date of clinical trial, whichever came first, assessed up to 4 weeks.
  The time from the start of treatment to the patient's recovery to Hughes Grade 2. The time from the start of protein A immunoadsorption or intravenous immunoglobulin treatment to the time the patient recovers to be able to walk independently for a distance of more than 5 meters.
Ventilator application time | For patients who require ventilator-assisted ventilation, from date of start use ventilator until participants leave the ventilator or end date of clinical trial, whichever came first, assessed up to 4 weeks.
  For patients with ventilator-assisted ventilation, the length of time from the beginning of treatment to leaving the ventilator.
Total time in ICU | From the date the patient enters the ICU until the patient leaves the ICU or the clinical trial ends, whichever came first, assessed up to 4 weeks.
  The total time that patients in the protein A immunoadsorption or intravenous immunoglobulin group were admitted to the ICU.
Changes of total lymphocyte count, interleukin-6, interleukin-8, cerebrospinal fluid protein | 2 weeks after starting treatment vs. baseline (before starting treatment)
  Compared with the results before treatment, changes of total lymphocyte count, interleukin-6, interleukin-8, cerebrospinal fluid protein after 2 weeks of the start of the treatment.
Changes of Compound muscle action potential and motor nerve conduction velocity of bilateral tibial nerves | 4 weeks after starting treatment vs. baseline (before starting treatment)
  Changes of Compound muscle action potential and motor nerve conduction velocity of bilateral tibial nerves before the treatment and 4 weeks after the start of the treatment in the protein A immunoadsorption or intravenous immunoglobulin group.

CONTACTS AND LOCATIONS:
Overall Officials: Junfang Teng, Prof, Study Director — The First Affiliated Hospital of Zhengzhou University; Wang Miao, Prof, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
After the clinical trial is completed, the individual participant data will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available after five years, permanent.
Access Criteria: No.